CLINICAL TRIAL: NCT02215330
Title: A Randomized, Double-masked, Placebo Controlled Study of the Beneficial Effects of Eplerenone on Central Serous Chorioretinopathy
Brief Title: A Study of the Beneficial Effects of Eplerenone on Central Serous Chorioretinopathy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prim. Univ-Prof. Dr. MBA, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPL; EK_14_170_0814 (Other: Ethikkommission der Stadt Wien)
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Central Serous Chorioretinopathy
Keywords: Central serous chorioretinopathy; Eplerenone; Photodynamic Therapy; Macula; Retina
MeSH Terms: conditions — Central Serous Chorioretinopathy | interventions — Eplerenone; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar pill (Placebo Comparator): Maltodextrin filled into capsules.
  1 Pill starting dosage
  Follow-up visits (every two weeks, beginning at week 4):
  * If subretinal fluid is present and the patient takes two pills a day dosage stays the same.
  * If no subretinal fluid is present, the patient will continue the present dosage for another 2 weeks and will then stop the medication.
  * If no subretinal fluid is present and the patient takes no medication everything stays the same.
  * If subretinal fluid is present again (recurrence) and the patient takes no medication, the medication will be re-started again, the patient has to take one tablet beginning at the following day
  Interventions: Drug: Maltodextrin
- Eplerenone (Experimental): Eplerenone 25mg pills triturated and filled into capsules.
  1 Pill starting dosage
  Follow-up visits (every two weeks, beginning at week 4):
  * If subretinal fluid is present and the patient takes two pills a day dosage stays the same.
  * If no subretinal fluid is present, the patient will continue the present dosage for another 2 weeks and will then stop the medication.
  * If no subretinal fluid is present and the patient takes no medication everything stays the same.
  * If subretinal fluid is present again (recurrence) and the patient takes no medication, the medication will be re-started again, the patient has to take one tablet beginning at the following day
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone
  Arms: Eplerenone
Drug: Maltodextrin
  Arms: Sugar pill

SUMMARY:
Central serous chorioretinopathy (CSC) is supposedly the fourth most common non-surgical retinopathy after age-related macular degeneration, diabetic retinopathy and branch retinal vein occlusion. The disease was first described by Albrecht von Graefe in 1866 as a 'recurrent central retinitis' and is nowadays commonly known as 'central serous chorioretinopathy', a term mainly coined by Donald Gass in the late 1960s.

Although the disease has been known for decades, the underlying mechanism is not yet fully understood. Numerous studies have shown an involvement of the retinal pigment epithelium (RPE) and the choroid which lead to accumulation of subretinal fluid with subsequent detachment of the neurosensory retina.

Among several assumed risk factors, high serum glucocorticoid levels seem to be related to the occurrence of CSC.

CSC typically affects young, male patients unilaterally and causes decreased and distorted vision, often associated with metamorphopsia, micropsia, dyschromatopsia and reduced contrast sensitivity. CSC can occur in an acute or chronic form. However, there is no agreement in the literature concerning the duration of the two forms. Some authors define CSC as chronic if there is persistent subretinal fluid for at least 6 months 11, others speak of chronic CSC when symptoms last longer than 3 months. In contrast there are studies where CSC is defined acute within the first 4 months. Spontaneously absorption is possible in up to 50% and normally leads to the recurrence of a normal visual acuity. Chronic CSC can result in a wide spread RPE damage and in a constantly reduction of visual acuity.

Structural changes in the retina and RPE have been found about 2 months after onset of the disease. Those changes can cause accumulation of photoreceptor outer segments, lead to consecutive atrophy of the photoreceptor cells and are associated with a loss of visual acuity.

Different concepts of treatment exist, but none of these may be deemed to be the golden standard. In the past few years several studies where CSC was treated with photodynamic therapy (PDT) or half-fluence PDT showed good visual outcomes and morphologic reconstitution. However, PDT is a destructive method which causes structural damage and can trigger other severe complications like choroidal ischemia and iatrogenic CNV. Furthermore, CSC is a self-limiting disease in many cases and physicians often hesitate to perform a relatively destructive therapeutical approach to treat a potentially self-limiting disease.

A newer, non-destructive therpeutical concept is the oral use of eplerenone a mineralocorticoid receptor antagonist. It is currently used in the treatment of hypertension and congestive heart failure. In the recent literature it was shown that eplerenone improved CSC and no serious adverse effects were observed in any case. However, no randomised controlled studies were performed comparing eplerenone with placebo to evaluate the clinical effect.

DETAILED DESCRIPTION:
Central serous chorioretinopathy (CSC) is supposedly the fourth most common non-surgical retinopathy after age-related macular degeneration, diabetic retinopathy and branch retinal vein occlusion. The disease was first described by Albrecht von Graefe in 1866 as a 'recurrent central retinitis' and is nowadays commonly known as 'central serous chorioretinopathy', a term mainly coined by Donald Gass in the late 1960s.

Although the disease has been known for decades, the underlying mechanism is not yet fully understood. Numerous studies have shown an involvement of the retinal pigment epithelium (RPE) and the choroid which lead to accumulation of subretinal fluid with subsequent detachment of the neurosensory retina.

Among several assumed risk factors, high serum glucocorticoid levels seem to be related to the occurrence of CSC.

CSC typically affects young, male patients unilaterally and causes decreased and distorted vision, often associated with metamorphopsia, micropsia, dyschromatopsia and reduced contrast sensitivity. CSC can occur in an acute or chronic form. However, there is no agreement in the literature concerning the duration of the two forms. Some authors define CSC as chronic if there is persistent subretinal fluid for at least 6 months 11, others speak of chronic CSC when symptoms last longer than 3 months. In contrast there are studies where CSC is defined acute within the first 4 months. Spontaneously absorption is possible in up to 50% and normally leads to the recurrence of a normal visual acuity. Chronic CSC can result in a wide spread RPE damage and in a constantly reduction of visual acuity.

Structural changes in the retina and RPE have been found about 2 months after onset of the disease. Those changes can cause accumulation of photoreceptor outer segments, lead to consecutive atrophy of the photoreceptor cells and are associated with a loss of visual acuity.

Different concepts of treatment exist, but none of these may be deemed to be the golden standard. In the past few years several studies where CSC was treated with photodynamic therapy (PDT) or half-fluence PDT showed good visual outcomes and morphologic reconstitution. However, PDT is a destructive method which causes structural damage and can trigger other severe complications like choroidal ischemia and iatrogenic CNV. Furthermore, CSC is a self-limiting disease in many cases and physicians often hesitate to perform a relatively destructive therapeutical approach to treat a potentially self-limiting disease.

A newer, non-destructive therpeutical concept is the oral use of eplerenone a mineralocorticoid receptor antagonist. It is currently used in the treatment of hypertension and congestive heart failure. In the recent literature it was shown that eplerenone improved CSC and no serious adverse effects were observed in any case. However, no randomised controlled studies were performed comparing eplerenone with placebo to evaluate the clinical effect.

Aim of this randomised controlled double-masked study is to compare the treatment effects of eplerenone versus placebo in patients with acute or chronic CSC with an untreated observational period of at least 2 months. If there is no sign of clinical improvement within the first 16 weeks after the onset of symptoms, patients will be offered half-fluence PDT.

In smaller case series, eplerenone was shown to be a valuable therapeutical option for patients suffering from CSC, but no randomised studies are available. The oral application was well tolerated by the patients and no severe side effects occurred.

The most common side effect of eplerenone is hyperkalemia making close monitoring in individuals with diabetes mellitus or renal disease necessary. In our study, blood tests according to the standard for eplerenone will be performed for all patients. Additionally, all patients in the study will be seen and examined by an internal medicine specialist sub-specialized in endocrinology prior to treatment and during the entire duration of the study.

Patients suffering from CSC included in this study will either receive eplerenone or placebo tablets. The treatment will start 2 months after recognition of first symptoms at the earliest. Therefore, patients with acute CSC are not missing out on treatment, as the usual "treatment" in this phase is observation only. Patients in the eplerenone group may benefit from taking part in this study, whereas patients in the control group will undergo the standard treatment (=observation only). Our current treatment protocol is to perform a half-fluence PDT approximately 4 months after onset of symptoms. All patients that do not improve within this time period will be offered to receive a half-fluence PDT. In the case of chronic CSC, with onset of symptoms or diagnosis more than 2 months of duration, eplerenone or placebo will nevertheless be offered with the above mentioned treatment period of 2 months and the rescue therapy option of half-fluence PDT in case of no signs of a positive treatment effect within 4 months of eplerenone therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from untreated CSC for less than two months
* Age 21 and older
* Written informed consent

Exclusion Criteria:

* Patients who have recently been treated with eplerenone
* Pregnancy or patients who are currently breast-feeding
* Patients who should not use eplerenone for any reason - an extensive internal medicine assessment will be performed in all patients prior to treatment start)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-03 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Difference in the number of successful treatments after 16 weeks, defined as complete absence of subretinal fluid on SD-OCT | 16 weeks
  Difference in the number of successful treatments after 16 weeks, defined as complete absence of subretinal fluid on SD-OCT, between the study and the control groups. The final evaluation will be performed by an external retina specialist. Significance testing will be performed using Fischer's exact test.

SECONDARY OUTCOMES:
Changes in visual acuity between eplerenone and placebo. | 16 weeks
Changes in retinal thickness between eplerenone and placebo. | 16 weeks
Changes in retinal volume between eplerenone and placebo. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, Prof, MBA, Principal Investigator — VIROS - Vienna Institute for Research in Ocular Surgers - Departement of Opthalmology - Hanusch Hospital Vienna, Vienna, Austria 1140
Locations (1):
- Oliver Findl, Vienna, Austria

REFERENCES:
- [Derived] Lange CA, Qureshi R, Pauleikhoff L. Interventions for central serous chorioretinopathy: a network meta-analysis. Cochrane Database Syst Rev. 2025 Jun 16;6(6):CD011841. doi: 10.1002/14651858.CD011841.pub3. PMID 40522203